CLINICAL TRIAL: NCT00385437
Title: Antidepressant Response to a Sedating Antidepressant Improves Driving Safety in Patients With Major Depressive Disorder
Brief Title: Sedating Antidepressant Improves Driving Safety in Patients With Major Depressive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Organon (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB-03-0255-A
Record Dates: First submitted 2006-10-05; First posted 2006-10-09 (Estimated); Last update posted 2006-10-09 (Estimated); Status verified 2006-02

CONDITIONS: Depression; Excessive Daytime Sleepiness
Keywords: Driving safety; maintenance of wakefulness test; major depressive disorder; mirtazapine
MeSH Terms: conditions — Depression; Disorders of Excessive Somnolence; Depressive Disorder, Major

INTERVENTIONS:
Behavioral: Driving Simulator Testing
Drug: Mirtazapine Treatment

SUMMARY:
This concurrent, two-part study will:

I) Using overnight sleep recordings, evaluate the short- and long-term sleep-promoting effects of the antidepressant mirtazapine (Remeron) in patients who have been prescribed this medication for major depressive disorder and sleep disruption.

II) Investigate the psychomotor performance of depressed patients using driving simulation testing before and during treatment with mitrazapine.

DETAILED DESCRIPTION:
In the treatment of depression, the role of sleep is important as there are mutual relationships between mood disorder and sleep disorders. Over 80% of major depressive disorder (MDD) patients report sleeping problems. Depression can strongly impair cognitive functioning and daytime alertness. (Mirtazapine (Remeron) is an antidepressant and sleep-promoting agent that has been available in Canada for a few years. However, research investigating the effects of mirtazapine on sleep is limited and it is not known what are the short- and long-term changes in sleep architecture associated with this drug and if daytime performance is affected.

Rationale:

The co-existence of depression and sleep difficulties are very common. Mirtazapine is marketed as a single modality of treatment for both depression and impaired sleep. As a sleep clinic in a psychiatry department, a single modality of treatment for depressive and sleep disorders is preferred by patients and can help improve compliance to treatment. However, there are only 7 published studies investigating the effects of mirtazapine and sleep and these have significant limitations. None of these studies have objectively examined mirtazapine's short- and long-term on sleep architecture and daytime function (daytime sleepiness, alertness, driving performance) in depressed patients. This study will address these issues.

Hypothesis:

I) Mirtazapine will produce both immediate and long- improvement effects on sleep in patients with major depressive disorders. There may be impairments in alertness for the first two days after starting treatment but daytime alertness will recover after one week.

II) Patients treated with mitrazapine will show a rapid, initial improvement in driving performance with recovery of sleep and slower, further improvement as treatment of their depression translates into better sleep quality as well as improvements in attention, alertness and concentration.

Study Design:

This pilot proposal is a two-part longitudinal, open-label clinical study with consecutive enrollment of subjects.

This research study will take place in conjunction with normal clinical practice. Patients with depression and sleep disorders are commonly seen in our sleep clinic and mirtazapine is one of several antidepressants that is prescribed by our clinicians. In this study, we will follow a group of patients who have been prescribed mirtazapine by one of our clinic physicians and who meet the inclusion and exclusion listed below. There will be an additional number of sleep studies (10 total versus the usual 2 or 3) performed; the usual daytime testing will be conducted as part of the standard of care (Multiple Sleep Latency Test (MSLT) and Maintenance of Wakefulness Test (MWT)); we will administer additional questionnaires to assess subjective sleepiness, alertness and fatigue; and, driving simulator testing will be conducted in accordance with our normal standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Fulfilling DSM-IV criteria for Major Depressive Disorder
* Score of Hamilton Rating Scale for Depression (HDRS-17) > 17
* Patient to be prescribed mirtazapine (Remeron) as determined by physician
* Subject has no known clinically significant abnormal vital signs or other clinical findings at screening.
* Patients should have a driving license for more than 3 years and drive over 15,000 km year.
* Females of childbearing potential must willingly use effective birth control.

Exclusion Criteria:

* Night shift workers.
* A history or present condition of: Bipolar Disorder or Depressive Disorder not Otherwise Specified,Schizophrenia or other psychotic disorders (according to DSM-IV), Schizotypal or Borderline personality disorder, Organic mental disorders
* A present condition of: Anxiety Disorders (according to DSM-IV), Eating Disorders, Postpartum Depression
* Epilepsy or a history of seizure disorder or ever received treatment with anticonvulsant medication for epilepsy or seizures
* PSG recording of an extremely abnormal sleep EEG (other than that which would be expected with depression)
* Alcohol or substance abuse (according to DSM-IV) during the last 6months prior to baseline.
* Any physical disease, which may explain the symptoms of depression.
* Any chronic physical disease, which is not stabilized.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16
Dates: Start 2003-04; Study Completion 2004-06

PRIMARY OUTCOMES:
Driving performance on the driving simulator

SECONDARY OUTCOMES:
Ability to maintain wakefulness

CONTACTS AND LOCATIONS:
Overall Officials: Colin M. Shapiro, MBBCh, PhD, Principal Investigator — University Health Network, Toronto; Sharon A. Chung, PhD, Study Director — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada

REFERENCES:
- [Background] Bulmash EL, Moller HJ, Kayumov L, Shen J, Wang X, Shapiro CM. Psychomotor disturbance in depression: assessment using a driving simulator paradigm. J Affect Disord. 2006 Jul;93(1-3):213-8. doi: 10.1016/j.jad.2006.01.015. Epub 2006 Mar 7. PMID 16522332
- [Result] Shen J, Chung SA, Kayumov L, Moller H, Hossain N, Wang X, Deb P, Sun F, Huang X, Novak M, Appleton D, Shapiro CM. Polysomnographic and symptomatological analyses of major depressive disorder patients treated with mirtazapine. Can J Psychiatry. 2006 Jan;51(1):27-34. doi: 10.1177/070674370605100106. PMID 16491981
- [Derived] Shen J, Moller HJ, Wang X, Chung SA, Shapiro GK, Li X, Shapiro CM. Mirtazapine, a sedating antidepressant, and improved driving safety in patients with major depressive disorder: a prospective, randomized trial of 28 patients. J Clin Psychiatry. 2009 Mar;70(3):370-7. doi: 10.4088/jcp.08m04234. Epub 2009 Jan 13. PMID 19192466